CLINICAL TRIAL: NCT02135406
Title: Pilot Study Of Redirected Autologous T Cells Engineered To Contain Anti-CD19 Attached To TCRζ And 4-1BB Signaling Domains Coupled With Salvage Autologous Stem-Cell Transplantation (ASCT) In Multiple Myeloma Patients With Early Relapse/Progression After Initial ASCT
Brief Title: CART-19 for Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC02413, 817462
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2018-02

CONDITIONS: Multiple Myeloma
Keywords: Adult; 18 years or older; multiple myeloma; poor prognosis; relapsed/progressive disease; within one year of first autologous stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multiple Myeloma Patients (Experimental): Adult subjects (18 years or older) with multiple myeloma and with poor prognosis by virtue of having relapsed/progressive disease within one year of first autologous stem cell transplantation.
  Interventions: Biological: CART-19 T cells

INTERVENTIONS:
Biological: CART-19 T cells

SUMMARY:
The primary goals: determine the safety, tolerability and engraftment potential of CART-19 T cells in patients undergoing salvage ASCT after early relapse following first ASCT. CART-19 cells transduced with a lentiviral vector to express anti-CD19 scFv TCR(zeta):41BB administered by intravenous infusion using a single infusion of 1-5x108 CART19-transduced T cells on day +2 after autologous stem cell infusion following high-dose melphalan.

ELIGIBILITY:
Inclusion Criteria - Subjects must have undergone a prior ASCT for MM and have progressed within 365 days of stem cell infusion. Patients who underwent syngeneic transplant (i.e., transplant from an identical twin donor) rather than autologous transplant are eligible and syngeneic transplant will be considered equivalent to ASCT for the purposes of these inclusion/exclusion criteria. Progression will be defined according to IMWG criteria for progressive disease143 (Table 4).

Subjects who have undergone two prior ASCTs as part of a planned tandem ASCT consolidation regimen are eligible.

Patients in whom first progression is identified between days 366 and 450 (inclusive) after ASCT will be eligible if progression is identified on their first evaluation for progression in this window and if they had not been evaluated between days 270 and 365 for progression. This clause is to account for practice patterns in which patients otherwise doing well are monitored infrequently (every 3-6 months) for relapse after they recover from their first ASCT. This will allow infrequently monitored patients to be included if progression is identified on their "12 month follow-up evaluation" if this appointment happens to be scheduled just outside the 365-day post-ASCT window. N.B.: There is no requirement that patients must enroll within 365 days of prior ASCT, and patients may be treated with other agents, including experimental agents, following relapse/progression after prior ASCT before enrollment on this study.

* Subjects must have received as part of their initial therapy for MM, prior to first ASCT, a regimen containing either bortezomib or lenalidomide.
* Subjects must have a confirmed diagnosis of active MM prior to first ASCT as defined by the IMWG criteria143, with the exception that patients treated for active MM on account of recurrent, complicated infections as the only clinical manifestation or on account of progressive smoldering MM with imminent clinical complications may be included.

Subjects must have signed written, informed consent. Subjects must be ≥ 18 and <70 years of age. Subjects must have an anticipated survival of >100 days after high-dose melphalan.

-Subjects must have adequate vital organ function as defined by the following criteria: Serum creatinine ≤ 2.5 or estimated creatinine clearance ≥30 ml/min and not dialysis-dependent.

Absolute neutrophil count ≥1000/μl and platelet count ≥50,000/μl. SGOT ≤ 3x the upper limit of normal and total bilirubin ≤ 2.0 mg/dl (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome).

Left ventricular ejection fraction (LVEF) ≥ 45% Adequate pulmonary function with FEV1, FVC, TLC, DLCO (after appropriate adjustment for lung volume and hemoglobin concentration) ≥40% of predicted values.

Toxicities from prior therapies must have recovered to grade ≤2 according to the CTC 4.0 criteria or to the subject's prior baseline.

* Subjects must have an ECOG performance status of 0-2, unless a higher performance status is due solely to bone pain.
* Subjects must be willing to comply with the requirements of the RevAssist program if maintenance lenalidomide is planned.
* Subjects must have measurable disease on study entry. Measurable disease may include quantifiable or detectable levels of serum or urine paraprotein. For patients with minimally secretory disease or non-secretory myeloma on study entry, serum free lambda or kappa light chain levels or the serum free light chain ratio may be measured and used for disease monitoring if abnormal. Likewise, for patients with IgA MM in which serum protein electrophoresis is deemed unreliable due to co-migration of normal serum proteins with the paraprotein, elevated total serum IgA levels may be considered measurable disease.
* Subjects must have stored in usable condition for second ASCT, as judged by the principal investigator, ≥3x106 CD34+ cells per kg of body weight (either autologous or syngeneic) stored in at least two bags such that after administration of the minimum dose of 2 x 106 CD34+ cells/kg required on this protocol that a separate aliquot of at least 1 x 106 CD34+ cells/kg remains for rescue infusion in the event of graft failure. Patients with inadequate stem cells stored may still sign consent and undergo a mobilization/collection procedure either before or after apheresis for T cell harvest. If this is required and is undertaken prior to apheresis for T cell harvest, two weeks must elapse between the last day of stem cell collection and apheresis for T cell harvest.

Table 5 IMWG Criteria for Progression

One or more of the following criteria must be met:

Increase of ≥25% from baseline in Serum M-component (the absolute increase must be ≥0.5 g/dl) (if baseline M-component is ≥5 g/dl, increases of ≥1 g/dl are sufficient to define progression) and/or Urine M-component (the absolute increase must be X200 mg/24 h ) and/or The difference between involved and uninvolved FLC levels (only in patients without measurable serum and urine M-protein levels) (the absolute increase must be >10 mg/dl).

Bone marrow plasma cell percentage (the absolute % must be ≥10%) For cases of IgA MM in which SPEPs are unavailable or are deemed unreliable due to migration of the paraprotein in the beta region, total IgA levels may be used to assess progression and response to therapy.

Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas.

Development of hypercalcemia (corrected serum calcium >11.5 mg/dl or 2.65 mmol/l) that can be attributed solely to the plasma cell proliferative disorder IMWG Criteria for Diagnosis of Multiple Myeloma Presence of an M-component in serum and/or urine plus clonal plasma cells in the bone marrow and/or a documented clonal plasmacytoma. In patients with no detectable M-component, an abnormal serum FLC ratio on the serum FLC assay can substitute and satisfy this criterion. For patients, with no serum or urine M-component and normal serum FLC ratio, the baseline bone marrow must have ≥10% clonal plasma cells; these patients are referred to as having 'non-secretory myeloma'. Patients with biopsy-proven amyloidosis and/or systemic light chain deposition disease (LCDD) should be classified as 'myeloma with documented amyloidosis' or 'myeloma with documented LCDD,' respectively if they have ≥30% plasma cells and/or myeloma-related bone disease.

PLUS one or more of the following, which must be attributable to the underlying plasma cell disorder:

Calcium elevation (>11.5 mg/dl) Renal insufficiency (creatinine >2 mg/dl) Anemia (hemoglobin <10 g/dl or at 2 g/dl below normal) Bone disease (lytic lesions or osteopenia)

Exclusion Criteria

Subjects must not:

* Be pregnant or lactating.
* Have inadequate venous access for or contraindications to leukapheresis.
* Have any active and uncontrolled infection.
* Have active or chronic hepatitis B [detectable hepatitis B surface antigen (HBsAg)], hepatitis C [positive serology (HCV Ab)], or HIV infection.
* Any uncontrolled medical disorder that would preclude participation as outlined.
* Have undergone allogeneic stem cell transplantation.
* Have received prior gene therapy or gene-modified cellular immunotherapy. Subject may have received, however, non-gene-modified autologous T-cells with their first ASCT in association with an anti-myeloma vaccine (e.g., hTERT or MAGEA3) or vaccination against infectious agents (e.g., influenza or pneumococcus) as was performed on our previous studies.
* Have undergone two prior ASCTs if the second ASCT was a salvage ASCT (defined as a second ASCT performed upon progression following first ASCT) rather than a second ASCT as part of a tandem ASCT consolidation regimen.
* Have auto-immune disease (including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis) that is active and severe in the judgment of the principal investigator, or have a history of autoimmune disease that has required prolonged immunosuppressive therapy in the judgment of the principal investigator.
* Have active central nervous system disease, including CNS involvement by malignancy or evidence of blood in the CNS such as subdural hematoma. If a subject has any neurological abnormality on examination, a baseline brain MRI is required to exclude structural disease and/or intracranial bleeding. Patients with clinically significant intracranial lesions should be excluded. Patients with common age-related changes that are not clinically significant (i.e. moderate small vessel ischemic changes) do not need to be excluded.
* Have a Class III/IV cardiovascular disability according to the New York Heart Association Classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward Stadtmauer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Garfall AL, Stadtmauer EA, Hwang WT, Lacey SF, Melenhorst JJ, Krevvata M, Carroll MP, Matsui WH, Wang Q, Dhodapkar MV, Dhodapkar K, Das R, Vogl DT, Weiss BM, Cohen AD, Mangan PA, Ayers EC, Nunez-Cruz S, Kulikovskaya I, Davis MM, Lamontagne A, Dengel K, Kerr ND, Young RM, Siegel DL, Levine BL, Milone MC, Maus MV, June CH. Anti-CD19 CAR T cells with high-dose melphalan and autologous stem cell transplantation for refractory multiple myeloma. JCI Insight. 2018 Apr 19;3(8):e120505. doi: 10.1172/jci.insight.120505. eCollection 2018 Apr 19. PMID 29669947
- [Derived] Garfall AL, Maus MV, Hwang WT, Lacey SF, Mahnke YD, Melenhorst JJ, Zheng Z, Vogl DT, Cohen AD, Weiss BM, Dengel K, Kerr ND, Bagg A, Levine BL, June CH, Stadtmauer EA. Chimeric Antigen Receptor T Cells against CD19 for Multiple Myeloma. N Engl J Med. 2015 Sep 10;373(11):1040-7. doi: 10.1056/NEJMoa1504542. PMID 26352815